CLINICAL TRIAL: NCT01657877
Title: In Situ Study to Confirm the Anti-caries Potential of a 1.1365% w/w Sodium Monofluorophosphate (1500ppm F) Dentifrice
Brief Title: Anti-caries Potential of a Sodium Monofluorophosphate and Calcium Sodium Phosphosilicate Dentifrice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RH01381
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CSP/SMFP Dentifrice (Experimental): Dentifrice containing high fluoride content as SMFP and CSP
  Interventions: Drug: Calcium sodium phosphosilicate; Drug: Sodium monoflurophosphate
- SMFP Dentifrice Prototype 1 (Active Comparator): Dentifrice containing high fluoride content as SMFP and no CSP
  Interventions: Drug: Sodium monoflurophosphate
- SMFP Dentifrice Prototype 2 (Active Comparator): Dentifrice containing low fluoride content as SMFP and no CSP
  Interventions: Drug: Sodium monoflurophosphate
- CSP Dentifrice (Active Comparator): Dentifrice containing CSP but no fluoride
  Interventions: Drug: Calcium sodium phosphosilicate
- Placebo Dentifrice (Placebo Comparator): Dentifrice containing no CSP and no fluoride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium sodium phosphosilicate — CSP high percentage weight by weight
  Arms: CSP Dentifrice; CSP/SMFP Dentifrice
Drug: Sodium monoflurophosphate — 500 to 1500 parts per million (ppm) of fluoride
  Arms: CSP/SMFP Dentifrice; SMFP Dentifrice Prototype 1; SMFP Dentifrice Prototype 2
Drug: Placebo — No CSP and no fluoride
  Arms: Placebo Dentifrice

SUMMARY:
In situ study to compare treatment effect on enamel remineralization potential, measured by surface microhardness recovery (SMHR) and Enamel Fluoride Uptake (EFU). The study will explore the efficacy of an experimental sodium monofluorophosphate (SMFP) dentifrice containing calcium sodium phosphosilicate (CSP) in comparison to an experimental SMFP only dentifrice.

ELIGIBILITY:
Inclusion Criteria:

* Wears a removable bilateral mandibular partial denture that has good stability and support, with sufficient room on each side in the posterior buccal flange area to accommodate two enamel specimens [required dimensions 12 x 7 millimeters (mm)].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one clinical site (US).
Pre-assignment Details: A total of 95 participants were screened, of which 79 were randomized. Of the subjects who were not randomized, 11 did not meet the study criteria; 3 had protocol violations; 2 withdrew consent.
Groups:
- Overall Participants: In this cross-over study, participant partial dentures were modified to hold two enamel specimens. Denture was modified at the start of the first treatment period to hold the enamel specimens. The participants were randomized using a computer generated program to receive following dentifrices:
  1. Dentifrice containing 1500 parts per million (ppm) as sodium monofluorophosphate (SMFP) + 5% calcium sodium phosphosilicate (CSP)
  2. Dentifrice containing 1500 ppm fluoride as SMFP + 0% CSP
  3. Dentifrice containing 500 ppm fluoride as SMFP + 0% CSP
  4. Dentifrice containing 0 ppm fluoride + 0% CSP
  5. Dentifrice containing 0 ppm fluoride + 5% CSP. The participants applied the given dentifrice as per their treatment group to a toothbrush and brushed their natural teeth twice daily for one timed minute. There was a washout period of 6 days between each treatment period.
Period: Overall Study
Arm/Group | Overall Participants
Started | 79
Received 500ppm Fluoride as SMFP+ 0% CSP | 70 (Discontinuations: 1 due to other reason in P2 and 1 protocol violation in P4)
Received 1500ppm Fluoride as SMFP+5% CSP | 75 (Discontinuations:2 withdrawal of consent in period (P) 1; 1 AE in P2;1 protocol violation in P3 & P4)
Received 0ppm Fluoride+ 5% CSP | 71 (Discontinuations: 1 protocol violation in P1 and P2 each and 1 withdrawal of consent in P1.)
Received 0ppm Fluoride+ 0% CSP | 69 (Discontinuation: 1 in P4 due to other reasons)
Received 1500ppm Fluoride as SMFP+0% CSP | 71 (Discontinuations: 1 protocol violation in P1 and 1 withdrawal of consent and AE in P3)
Completed | 65
Not Completed | 14
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 6
Not completed — Adverse Event | 2
Not completed — Other Reason | 2

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline characteristics.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 33

OUTCOME MEASURES:

1. Secondary Outcome: Percentage (%) Change in SMH Following 21 Days of Twice Daily Treatment With 500 Ppm Fluoride as SMFP and 0 % CSP Dentifrice, 0 Ppm Fluoride and 0% CSP, and 0 Ppm Fluoride and 5 % CSP.
Description: Percent SMH recovery (SMHR) was calculated from hardness values of enamel specimens at baseline (B), after in-situ hardening (R) and after first demineralization challenge (D1) using formula: [(D1-R)/ (D1-B)]*100. A greater percentage change in SMHR represents a better remineralisation and hence a better outcome.
Time Frame: Baseline to 21 days
Population: PP population:all randomized participants in the ITT population who had no protocol violations leading to exclusion of all efficacy data from analyses.
Measure: Mean (Standard Error); unit: Percentage SMHR
Groups:
- Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 500 ppm fluoride as SMFP and 0 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 0 Ppm Fluoride + 0% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 0 ppm fluoride and 0 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 0 Ppm Fluoride + 5% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 0 ppm fluoride and 5 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
Arm/Group | Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 5% CSP
Number analyzed (Participants) | 70 | 69 | 70
Percentage SMHR | 18.72 (1.649) | 14.74 (1.362) | 14.01 (1.392)

2. Secondary Outcome: Enamel Fluoride Uptake (EFU)
Description: Change to EFU was determine using a microdrill enamel biopsy of the in situ enamel specimens.
Time Frame: Baseline to 21 days
Population: PP population: all randomized participants in the ITT population who had no protocol violations leading to exclusion of all efficacy data from analyses. Missing data was not imputed. Due to drop out there were differences in the number of participants analyzed per treatment group.
Measure: Mean (Standard Error); unit: ppm EFU
Groups:
- Dentifrice Containing 1500 Ppm Fluoride as SMFP + 5% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 1500 ppm fluoride as SMFP and 5 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 1500 Ppm Fluoride as SMFP + 0% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 1500 ppm fluoride as SMFP and 0 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 0 Ppm Fluoride + 0% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing no fluoride and no CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 0 Ppm Fluoride + 5% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing no fluoride and 5 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
Arm/Group | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 5% CSP | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 5% CSP
Number analyzed (Participants) | 75 | 70 | 70 | 69 | 70
ppm EFU | 15.58 (0.784) | 14.85 (0.729) | 9.23 (0.440) | 4.17 (0.241) | 4.54 (0.291)

3. Primary Outcome: Percentage (%) Change in Surface Microhardness (SMH) Following 21 Days of Twice Daily Treatment With the 1500 Ppm Fluoride + 5% CSP Dentifrice and With the 1500 Ppm Fluoride Dentifrice.
Description: as for outcome 1
Time Frame: Baseline to 21 days
Population: Per protocol (PP) population: The per protocol (PP) population was defined as those subjects in the intention to treat population who did not have protocol violations leading to exclusion of all efficacy data from analyses. Missing data was not imputed.
Measure: Mean (Standard Error); unit: Percentage SMHR
Groups:
- Dentifrice Containing 1500ppm Fluoride as SMFP + 0% CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 1500 ppm fluoride as SMFP and 0 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
- Dentifrice Containing 1500ppm Fluoride as SMFP + 5 % CSP: Participants applied a full ribbon of the dentifrice (approximately 1.5 g) containing 1500 ppm fluoride as SMFP and 5 % CSP, to a toothbrush and brushed their natural teeth twice daily for one timed minute.
Arm/Group | Dentifrice Containing 1500ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 1500ppm Fluoride as SMFP + 5 % CSP
Number analyzed (Participants) | 70 | 75
Percentage SMHR | 30.15 (2.447) | 32.32 (2.673)
Statistical Analysis 1: Comparison: Dentifrice Containing 1500ppm Fluoride as SMFP + 0% CSP vs Dentifrice Containing 1500ppm Fluoride as SMFP + 5 % CSP; The null hypothesis states that the population mean for the 1500 ppm fluoride as SMFP + 0% CSP minus the population mean for the 1500 ppm fluoride as SMFP and 5% CSP dentifrice is more than 6 %; Test type: Non-Inferiority or Equivalence — The success criterion for this study was to observe the upper bound of the 2-sided 95% confidence interval for difference in % change in SMHR to be <= 6 units SMHR i.e. 1500 ppm fluoride as SMFP + 5% CSP is no more than 6 units inferior to the 1500 ppm fluoride as SMFP + 0 % CSP dentifrice; p = 0.2601, ANOVA; Based on the mixed effects ANOVA considering treatment and study period as factors, and subject as random effect; Adjusted mean difference = -2.23, 95% CI 2-sided [-6.11 to 1.66] — Difference is 1500 ppm fluoride as SMFP and 0 % CSP minus 1500 ppm fluoride as SMFP and 5 % CSP such that a positive difference favors 1500 ppm fluoride as SMFP and 0 % CSP

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the investigational product (or washout product), and until 5 days following last administration of the investigational product.
Arm/Group | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 5% CSP | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 0% CSP | Dentifrice Containing 0 Ppm Fluoride + 5% CSP
Serious Adverse Events (participants affected / at risk) | 1/75 | 0/71 | 2/70 | 0/69 | 0/71
Other Adverse Events (participants affected / at risk) | 18/75 | 13/71 | 14/70 | 11/69 | 13/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 5% CSP (N=75) | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 0% CSP (N=71) | Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP (N=70) | Dentifrice Containing 0 Ppm Fluoride + 0% CSP (N=69) | Dentifrice Containing 0 Ppm Fluoride + 5% CSP (N=71)
Invasive lobular carcinoma of left breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unstable angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple myeloma of bones (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 5% CSP (N=75) | Dentifrice Containing 1500 Ppm Fluoride as SMFP + 0% CSP (N=71) | Dentifrice Containing 500 Ppm Fluoride as SMFP + 0% CSP (N=70) | Dentifrice Containing 0 Ppm Fluoride + 0% CSP (N=69) | Dentifrice Containing 0 Ppm Fluoride + 5% CSP (N=71)
Gingival erythema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental caries (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth repair (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.